CLINICAL TRIAL: NCT00886509
Title: Subcutaneous Administration of Pegylated Granulocyte-Colony Stimulating Factor for Long-Term Promotion of Collateral Growth in Patients With Coronary Artery Disease
Brief Title: Peg-Granulocyte-Colony Stimulating Factor (GCSF) for Coronary Collateral Growth in Coronary Artery Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 199/2008
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Stable; Coronary Collaterals; Therapeutic Collateral Promotion (TCP)
MeSH Terms: conditions — Coronary Artery Disease | interventions — pegfilgrastim; pegylated granulocyte colony-stimulating factor, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collateral promotion; PCI after 6 months (Experimental): First pegGCSF or placebo; PCI after 6 months
  Interventions: Biological: pegfilgrastim; Other: Placebo
- Collateral promotion after PCI at baseline (Experimental): Collateral promotion with pegGCSF after PCI at baseline
  Interventions: Biological: pegfilgrastim

INTERVENTIONS:
Biological: pegfilgrastim — s.c. administration of pegylated G-CSF over 6 months
  Other Names: Peg-GCSF; Peg-G-CSF; PEG-rmetHuG-CSF; Amgen brand of pegfilgrastim; Neulasta; pegylated (r-G-CSF)
Other: Placebo — Placebo control Arm 1: Collateral promotion; PCI after 6 months
  Other Names: Placebo control
  Arms: Collateral promotion; PCI after 6 months

SUMMARY:
The purpose of this study in patients with stable coronary artery disease (CAD) treatable by PCI (percutaneous coronary intervention) is to evaluate the long-term efficacy and safety of subcutaneously applied, pegylated granulocyte colony stimulating factor (Pegfilgrastim, PEG-G-CSF; Neulasta®, Amgen Switzerland) with regard to the promotion of collateral growth.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death in industrialized countries. Current revascularization therapies are PCI or surgical revascularization. However, inherent to them are procedure-related risks and the fact, that progression of CAD is not prevented. Additionally, up to one fourth of all CAD patients are not amenable to standard revascularization therapies. Thus, there is a need for alternative therapies. The coronary collateral circulation is prevalent in humans, and in CAD the amount of collateral flow is a pivotal protective factor with respect to infarct size, all-cause- and cardiac mortality. Coronary collateral growth promotion is an alternative to conventional revascularization which can be achieved by cytokine-based approaches (e.g. with colony-stimulating factor-therapy) in humans. The goal of collateral promotion is to reduce myocardial damage in case of a coronary occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. 1- to 3-vessel coronary artery disease (CAD)
3. Stable angina pectoris
4. At least 1 stenotic lesion suitable for PCI
5. No Q-wave myocardial infarction in the area undergoing CFI measurement
6. Written informed consent to participate in the study

Exclusion Criteria:

1. Acute myocardial infarction
2. Unstable CAD
3. CAD treated best by CABG
4. Patients with overt neoplastic disease
5. Patients with diabetic retinopathy
6. Liver or kidney disease
7. Pre-menopausal women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Collateral flow index (CFI) | 6 months

SECONDARY OUTCOMES:
Myocardial blood flow (MBF) during hyperemia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD, Prof., Study Chair — University of Bern; Tobias Traupe, MD, Principal Investigator — University Hospital Berne; Michael Stoller, MD, Principal Investigator — University Hospital Berne
Locations (2):
- Switzerland (2):
  - University Hospital Berne, Bern, Canton of Bern
  - University Hospital Berne, Bern

REFERENCES:
- [Background] Meier P, Gloekler S, de Marchi SF, Indermuehle A, Rutz T, Traupe T, Steck H, Vogel R, Seiler C. Myocardial salvage through coronary collateral growth by granulocyte colony-stimulating factor in chronic coronary artery disease: a controlled randomized trial. Circulation. 2009 Oct 6;120(14):1355-63. doi: 10.1161/CIRCULATIONAHA.109.866269. Epub 2009 Sep 21. PMID 19770393